CLINICAL TRIAL: NCT02993133
Title: Pharmacokinetics Study of Mycophenolic Acid in Patients With an Autoimmune Bullous Dermatose, Pemphigus or Cicatricial Pemphigoid.
Acronym: PEMPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I14027 / PEMPA
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2018-06

CONDITIONS: Autoimmune Bullous Dermatose
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 60 patients will be used to build and validate the system (Experimental): The first 30 patients will be used to build and validate the pharmacokinetic modeling of MPA in pemphigus.The 30 patients included later will provide additional data.
  Interventions: Drug: Cellcept® in autoimmune bullous dermatoses

INTERVENTIONS:
Drug: Cellcept® in autoimmune bullous dermatoses — The administration will follow the recommendations for the use of Cellcept® in autoimmune bullous dermatoses

SUMMARY:
The main autoimmune bullous dermatoses are pemphigus and cicatricial pemphigoid. Pemphigus is an autoimmune dermatological disease characterized by the production of anti-desmoclesin antibodies 1 and 3, affecting the skin and mucous membranes.The cicatricial pemphigoid is an autoimmune dermatological disease, characterized by the production of anti-zone antibodies of the basal membrane and characterized by a predominant mucosal involvement. Mycophenolic acid (MPA) is an increasingly used form of corticosteroid. Despite its increasing use, pharmacokinetics in autoimmune bullous dermatosis remain little studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years.
* Patient treated by Mycophénolate Mofétil (MMF) per os (Cellcept®) for an autoimmune bullous dermatose (pemphigus or cicatricial pemphigoid) for at least 30 days according to the recommendations (PNDS Pemphigus and cicatricial pemphigoid HAS 2011)
* Patient able to understand the nature, purpose and methodology of the study
* Patient affiliated to the French social security system or equivalent
* Patient who have signed an informed consent form

Exclusion Criteria:

* Pregnant or breast-feeding women or women of childbearing potential without efficient contraception (based on a declaration)
* Patient under legal protection.
* Patient deprived of freedom
* Patient with any altered mental status or any psychiatric condition that would interfere with the understanding of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Bayesian estimator performance | 8 hours
  The evaluation of the Bayesian estimator performance will be based on its capacity to predict MPA AUC (Area Under the Curve), expressed as the bias (%) and the precision (root mean square error; RMSE) between the predicted AUC calculated using a limited number of samples performed in the first 4 hours post dosing and the observed AUC estimated using the reference method (trapezoidal rule method). A Bland Altman curve will be constructed.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Avicenne - AP-HP, Paris
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No